CLINICAL TRIAL: NCT07316595
Title: A Clinical Study of the Efficacy and Safety of Conditioning With Low Doses of Treosulfan Before Allogeneic Hematopoietic Stem Cell Transplantation for Patients With Nijmegen Breakage Syndrome
Brief Title: Study of Treosulfan-Based Conditioning for HSCT in Nijmegen Breakage Syndrome
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Collaborators: Russian Children's Clinical Hospital of the N.I. Pirogov Russian National Research Medical University (Unknown); Regional Children's Clinical Hospital, Yekaterinburg (Unknown); Morozov Children's Municipal Clinical Hospital of the Moscow City Health Department State-Financed H (Other Government); Raisa Gorbacheva Memorial Research Institute for Pediatric Oncology, Hematology and Transplantation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCHPOI- 2025-9
Record Dates: First submitted 2025-11-20; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: HSCT; Nijmegen Breakage Syndrome; Treosulfan Based Conditioning
MeSH Terms: conditions — Nijmegen Breakage Syndrome | interventions — treosulfan

STUDY DESIGN:
Intervention Model Description: We are planning a study to investigate treosulfan-based conditioning in patients with Nijmegen breakage syndrome, which will stratify patients based on the presence or absence of malignant disease. Patients without a tumor will receive treosulfan at a dose of 21 g/m², and patients with a tumor will receive 30 g/m².
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with Nijmegen breakage syndrome without malignant disease. (Active Comparator)
  Interventions: Drug: Treosulfan (Treo)
- Patients with Nijmegen breakage syndrome and malignant disease. (Active Comparator)
  Interventions: Drug: Treosulfan (Treo)

INTERVENTIONS:
Drug: Treosulfan (Treo) — We are planning a multicenter study to investigate treosulfan-based conditioning in patients with Nijmegen breakage syndrome, which will stratify patients based on the presence or absence of malignant disease. Patients without a tumor will receive treosulfan at a dose of 21 g/m², and patients with a tumor will receive 30 g/m²

SUMMARY:
Nijmegen breakage syndrome is one of the DNA repair defect disorders. A characteristic feature of these syndromes is a predisposition to the development of malignant neoplasms. The only curative option for the combined immunodeficiency in Nijmegen breakage syndrome is allogeneic hematopoietic stem cell transplantation (HSCT). In addition to correcting the immunodeficiency, HSCT can reduce the risk of developing hematopoietic tumors.

Due to the increased sensitivity of cells in patients with Nijmegen breakage syndrome to alkylating drugs, the use of standard myeloablative conditioning regimens for this disease significantly increases the risks of toxic complications and transplant-related mortality.

Treosulfan is an alkylating agent that has demonstrated efficacy with comparatively low risks of toxic complications when used as part of conditioning prior to allogeneic HSCT for various diseases in patients of all age groups. There is currently experience using treosulfan in patients with Nijmegen breakage syndrome at reduced doses (21 and 30 g/m²). However, a number of questions remain unresolved. Based on our previous experience, a dose of 21 g/m² is sufficient for patients with Nijmegen breakage syndrome without a malignant disease, as it ensures good graft function (a high probability of full donor chimerism and control of the immunodeficiency). At the same time, there is reason to believe that this dose is insufficient to provide an antitumor effect from the conditioning.

We are planning a multicenter study to investigate treosulfan-based conditioning in patients with Nijmegen breakage syndrome, which will stratify patients based on the presence or absence of malignant disease. Patients without a tumor will receive treosulfan at a dose of 21 g/m², and patients with a tumor will receive 30 g/m².

ELIGIBILITY:
Inclusion Criteria:

* genetically confirmed Nijmegen breakage syndrome
* availability of informed consent for study participation, signed by the patient (ages 14 to 21) and/or their legal representative (ages 0 to 18).
* absence of contraindications to HSCT based on the patient's somatic status.

Exclusion Criteria:

* other DNA repair deficiency syndromes (both specified and unspecified)

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate event-free survival (EFS), defined by the occurrence of death, graft rejection, or development of secondary malignancy/relapse. | 2 years
  Event-free survival in patients with Nijmegen syndrome is the primary criterion for assessing the effectiveness of HSCT. It was precisely the need to solve the problems of graft rejection, relapses of malignant diseases, and secondary tumors that became the main reasons for initiating this study.

SECONDARY OUTCOMES:
Overall survival | 2 years
To evaluate the rate of transplant-associated mortality. | 2 years
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | 3 months
Probability of graft rejection | 2 years
Frequency of Complete Donor and Mixed Chimerism after HSCT | 1 year
Incidence of acute GVHD. | 1 year
Incidence of chronic GVHD. | 2 years
To assess the kinetics of immune reconstitution | 1 year

IPD SHARING:
Plan to Share IPD: No